CLINICAL TRIAL: NCT00627094
Title: A Randomised, Controlled and Double-blind Clinical Investigation on the Effectiveness and Safety of a Foam Dressing Biatain Ibu Non-adhesive vs. Biatain Non-adhesive, in Painful Chronic Venous Leg Ulcers
Brief Title: Biatain Ibu vs. Biatain in Painful Chronic Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DK143WS
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Leg Ulcers
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biatain Ibu (Experimental): Biatain Ibu
  Interventions: Device: Biatain Ibu
- Biatain (Active Comparator): Biatain
  Interventions: Device: Biatain

INTERVENTIONS:
Device: Biatain — A standard polyurethane foam dressing Biatain non-adhesive (Coloplast A/S) with an elastic semi-permeable backing film, size 15x15 cm. The product is CE marked.
  Other Names: Coloplast Biatain
  Arms: Biatain
Device: Biatain Ibu — Biatain Ibu non-adhesive (Coloplast A/S), a polyurethane foam dressing with an elastic semi-permeable backing film with an added pain relieving medicinal substance ibuprofen (Albermarle Inc.), size 15x15 cm. The product is CE marked.
  Other Names: Coloplast Biatain-Ibu
  Arms: Biatain Ibu

SUMMARY:
The objective of this investigation is to demonstrate the effectiveness and safety of Biatain Ibu non-adhesive foam dressing compared to Biatain non-adhesive foam dressing.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Chronic venous leg ulcer on the lower leg
* Ulcer duration >= 8 weeks
* Pain intensity in study ulcer at least 4 on an 11-point numerical box scale (NBS): 0= no pain, 10= worst possible pain
* Exudate level moderate to high
* Ulcer size min 1.6 cm and max 11 cm in any direction
* Ankle/brachial index >= 0.8
* Treated with moist wound healing during the past 2 weeks prior to inclusion
* Adequate compression therapy during the past 2 weeks prior to inclusion
* The patient is cognitive capable of evaluating his/her pain relief and pain intensity
* The patient is able to understand the treatment and is willing to comply with the treatment regimen.
* The patient is able to complete the patient diary
* The patient is willing and able to give written informed consent

Exclusion Criteria:

* Painful ulcers that have been treatment resistant to analgesics for the past 6 months or more
* Pregnant or lactating women
* Known and verified hypersensitivity to any content of the products used in this investigation
* Local infection (bacterial imbalanced wound) in the study ulcer
* Clinical infection in the study ulcer
* Diseases: Vasculitis, erysipelas and cellulitis of the peri-ulcer skin
* The investigator considers the patient not eligible
* Diseases and conditions where ibuprofen or other analgesics are contraindicated (including known hypersensitivity to Aspirin (acetylsalicylic acid) or other analgesics, especially associated with a history of asthma, rhinitis or urticaria)
* Diabetes
* Use of per need medication for the past 3 days
* Concomitant treatment with systemic antibiotics other than nitrofurantoin
* Concomitant treatment with systemic corticosteroids (more than 10 mg/day prednisolon or equivalent) or other immunosuppressants within 1 month prior to inclusion
* Concomitant treatment with cancer chemotherapeutics
* Concomitant participation in other studies
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Fogh, MD, Principal Investigator — Aarhus University Hospital
Locations (13):
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Odense Universitets Hospital, Odense
- France (2):
  - CHU de Brest, Arras
  - CHU de Nancy - Hôpital Fournier, Nancy
- Germany (6):
  - Department for Dermatology, University School of Medicine, Essen
  - Georg-August-Universität Göttingen, Göttingen
  - Klinik für Dermatologie und Venerologie, Hanover
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Dr. Renzo Bause Praxis, Lüdenscheid
  - Fachartzpraxis für Dermatologie, Allergologie, Lasermedizin, Mahlow
- Spain (2):
  - C.S. SERGAS Rosalía de Castro - Enfermero, Vigo, Pontevedra
  - Hospital de Fuenlabrada, Fuenlabrada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Biatain Ibu: Biatain foam dressing containing Ibuprofen
- Biatain: Biatain Foam dressing without ibuprofen - control
Period: Overall Study
Arm/Group | Biatain Ibu | Biatain
Started | 60 | 60
Completed | 48 | 45
Not Completed | 12 | 15
Not completed — Adverse Event | 8 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — ulcer healed | 1 | 7
Not completed — Other reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biatain Ibu | Biatain | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: YEARS]
  Age | 71.6 (12.8) | 69.5 (12.5) | 70.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 82
  Male | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  France | 3 | 3 | 6
  Spain | 3 | 3 | 6
  Denmark | 32 | 32 | 64
  Germany | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief
Description: The distribution of pain relief assesment during day 1 to 5. The pain relief was registrated on 5-point verbal rating scales (evening/morning) from day 1 to day 5 after start of treatment.
Time Frame: Pain relief (morning/evening) after start of treatment from day 1 (evening) to day 5 (morning)
Population: ITT population
Measure: Number; unit: percentage of scores within category
Units Other Than Participants: Total Number of scores day 1-5
Arm/Group | Biatain Ibu | Biatain
Number analyzed (Participants) | 59 | 59
Number analyzed (Total Number of scores day 1-5) | 468 | 463
percentage of scores within category
  No Pain Relief | 22 | 31
  Slight Pain Relief | 26 | 31
  Moderate Pain Relief | 30 | 26
  A lot Pain Relief | 19 | 11
  Complete Pain Relief | 3 | 1
Statistical Analysis 1: Comparison: Biatain Ibu vs Biatain; The null hypothesis to be tested was that the distributions of categorical responses were the same; Test type: Superiority or Other; p = 0.0438, Chi-squared — In order to obtain 90% power to show superiority of Biatain Ibu compared to Biatain, a sample size of 60 pts per group (assuming a 15% drop-out rate) was found by simulating data from multi-nomial distributions over time; Result based on ITT population (evening). PP-analysis show a strong tendency (not significant) in favour of Biatain Ibu supporting the ITT-analysis; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.02 to 2.96]

2. Secondary Outcome: Pain Intensity (PI) Change
Description: Pain intensity (PI) assesment performed daily during the days 1-5. Pain intensity assesment performed on a 11 point numerical box scale: 0 was no pain and 10 was worst possible pain. A positive outcome measure value (PI (baseline) - PI (day 4 evening)) means that PI has decreased since baseline and thus reflects clinical improvement (patients suffer less from pain).
Time Frame: Change from baseline in Pain Intensity (PI) on day 4 evening
Population: PP-population (The PP population consisted of all randomized subjects that fulfilled the inclusion/exclusion criteria and which did not violate the protocol in a serious way day 1-5) - Evaluation performed on un-blinded data before database lock.
Measure: Mean (Standard Deviation); unit: Change in PI since baseline
Arm/Group | Biatain Ibu | Biatain
Number analyzed (Participants) | 60 | 60
Change in PI since baseline | 2.2 (2.2) | 1.9 (2.4)

3. Secondary Outcome: Change From Baseline in Ulcer Area
Description: Relative change from baseline in ulcer area using last observation carried forward. A positive outcome value Means that wound size has decreased and thus reflects wound healing (clinical improvement)
Time Frame: Change from baseline to end of trial (day 43)
Population: ITT population
Measure: Median (Standard Deviation); unit: Relative change from baseline in percent
Arm/Group | Biatain Ibu | Biatain
Number analyzed (Participants) | 60 | 60
Relative change from baseline in percent | 59 (82) | 50 (60)

4. Secondary Outcome: Adverse Events
Description: Number of Adverse events reported which were evaluated to be related or possible related to the device
Time Frame: Continuously from start of treatment to end of trial (day 43)
Measure: Number; unit: Number of AE
Arm/Group | Biatain Ibu | Biatain
Number analyzed (Participants) | 60 | 60
Number of AE | 4 | 6

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Biatain: Biatain foam dressing without ibuprofen
Arm/Group | Biatain Ibu | Biatain
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/60
Other Adverse Events (participants affected / at risk) | 4/60 | 6/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biatain Ibu (N=60) | Biatain (N=60)
Hospitalisation due to gastritis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biatain Ibu (N=60) | Biatain (N=60)
Contact dermatitis in the peri-ulcer skin (Skin and subcutaneous tissue disorders) | 1 | 4
Increased pain in study ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Blisters at the edge of the dressing (Skin and subcutaneous tissue disorders) | 1 | 0
Infection in study ulcer (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less